CLINICAL TRIAL: NCT07298798
Title: Comparison of the Closed Kinetic Chain and Isometric Exercise in Female Patient With Patellofemoral Pain Syndrome Associated With Knee Osteoarthritis: A Randomized Control Trial
Brief Title: To Compare the Effect of Closed Kinetic Chain and Isometric Exercises in Reducing Pain and Improving Functional Disability in Patients With Patellofemoral Pain Syndrome Associated With Knee Osteoarthritis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, FAKHRA ASGHAR, Principal Investigator, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB4014/DUHS/Approval/2025/268
Record Dates: First submitted 2025-08-26; First posted 2025-12-23 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Experimental: GroupA .will be give treatment closed kinetic chain exercise i.e Terminal knee extension and VMO squat.
  GroupB .will be give treatment isometric exercise i.e SLR and Static quads.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GroupA . given treatment closed kinetic chain exercise (Experimental): Terminal knee extension, The patient stand facing the plinth with feet shoulder-width apart and a theraband looped around their knee and other plinth legs. patient bend their knees to a 30-degree angle, extend their leg against the band's resistance, and hold this position for six seconds.
  VMO squat, The position of patient, hip and knee will bend, weight of the body on feet and feet about shoulder width apart and turn the feet outward about 45 degrees and position hold for 30 second.
  Interventions: Behavioral: Terminal knee extension. .VMO squat. [TheraBand]
- GroupB . given treatment isometric exercise SLR, Static quads. (Experimental): Static Quads The patient is long sitting or supine on their back, with a foam roll or towel behind their knee. Contract your quadriceps muscles while pressing down on the towel, maintaining this position for five seconds.
  Straight leg raising (SLR) The patient will be laying in supine, and before the exercise's lifting phase, a maximal isometric quadriceps contraction will be executed, followed by raising the leg to a height of 10cm above the plinth for 10 seconds.
  Interventions: Behavioral: Isometric exercises [knee roller]

INTERVENTIONS:
Behavioral: Terminal knee extension. .VMO squat. [TheraBand] — Terminal knee extension, The patient stand facing the plinth with feet shoulder-width apart and a theraband looped around their knee and other plinth legs. They bend their knees to a 30-degree angle, extend their leg against the band's resistance, and hold this position for six seconds.
  VMO squat, The position of patient, hip and knee will bend, weight of the body on feet and feet about shoulder width apart and turnthe feet outward about 45 degrees and position hold for 30 second.
  Arms: GroupA . given treatment closed kinetic chain exercise
Behavioral: Isometric exercises [knee roller] — Static Quads The patient is long sitting or supine on their back, with a foam roll or towel behind their knee.
  Contract your quadriceps muscles while pressing down on the towel, maintaining this position for five seconds. Straight leg raising (SLR) The patient will be laying in supine, and before the exercise's lifting phase, a maximal isometric quadriceps contraction will be executed, followed by raising the leg to a height of 10 cm above the plinth for 10 seconds.
  Arms: GroupB . given treatment isometric exercise SLR, Static quads.

SUMMARY:
Investigator study aims to compare the benefits of isometric exercise and closed kinetic chain exercises in strengthening programs to lessen pain along with enhance functionality in patients with PFP that are being associated with osteoarthritis and the assessment of PFP pertains to its recognition and the determination of significant therapeutic techniques. 70 Participants from the department of physiotherapy, Civil Hospital Karachi CHK and Dow University of Health Science (DIPMR) will be randomly assigned into two groups, an experimental group receiving closed kinetic chain exercise, and a control group receiving isometric exercises. The therapy will last four weeks, consisting of twelfth sessions. There will be 35 to 40 minutes in each session, Patients will be evaluated on primary outcome measure, pain intensity and functional limitation using various scales, including the numerical pain rating scale (NPRS) and Kujala/anterior knee pain scale (AKPS)

DETAILED DESCRIPTION:
The most prevalent issue of musculoskeletal knee joint that impact is patellofemoral pain syndrome (PFPS) particularly in young adults and the elderly, causing severe discomfort behind and around the patella, making it the primary etiology for anterior knee discomfort. Patellofemoral joint may be the first compartment affected in early knee osteoarthritis. Most exercise programs designed for treating p a t e l l o f e m o r a l p a i n ( PFP) focus on strengthening the quadriceps, primarily the vastus medialis oblique (VMO). A rehabilitation program including closed kinetic chain exercises and isometric exercises may be beneficial for patients with patellofemoral pain (PFP) to improve their functional limitations and minimize pain. Closed kinetic chain exercises improve functional movement patterns, while isometric exercises are better tolerated during pain or inflammation. The effectiveness of these approaches in individuals with patellofemoral pain (PFP) associated with knee OA is unclear, but understanding their differential impacts can guide targeted rehabilitation strategies for this complex patient population. Investigator aims to compare the benefits of isometric exercise and closed kinetic chain exercises in strengthening programs to lessen pain along with enhance functionality in patients with PFP that are being associated with osteoarthritis, Participants from the department of physiotherapy, Civil Hospital Karachi CHK and Dow University of Health Science (DIPMR) will be randomly assigned into two groups, an experimental group receiving closed kinetic chain exercise, and a control group receiving isometric exercises. The therapy will last four weeks, consisting of twelfth sessions. There will be 35 to 40 minutes in each session, Patients will be evaluated on pain intensity and functional limitation using various scales, including the numerical pain rating scale (NPRS) and Kujala/anterior knee pain scale (AKPS).

ELIGIBILITY:
Inclusion Criteria

* Age between (35 to 60) years.
* Gender: female.
* The numerical pain rating scale (NPRS) is greater than three out often i.e. 3/10 score.
* Patient experiences anterior knee pain due to such activities like squatting, prolonged sitting, running and stair climbing.
* Patient with unilateral or bilateral knee pain with positive radiographic imaging.
* Patients have grade 1 and 2 knee osteoarthritis (K&L classification).

Exclusion Criteria

* Any past record of knee surgery.
* Any past record of knee fracture.
* Patients with any neurological disorder.
* Cancer, malignancy or any bone tumor.
* Comorbid like diabetes mellitus.
* Any systemic inflammatory arthritis.

Ages: 35 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 70 (Actual)
Dates: Start 2023-11-09 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2027-11-08 (Estimated)

PRIMARY OUTCOMES:
numerical pain rating scale (NPRS) | 12th sessions for four weeks ,outcome measures will take place both, at the baseline when intervention start and four weeks, following the intervention
  1. Numerical pain rating scale (NPRS) Pain intensity will measure using NPR scale (no need for permission), a reliable instrument retest reliability of 0.95 , 0 represents no pain and 10 represents severe suffering.
  10= indicate worse pain 5= indicate moderate pain 0 = indicate no pain.
. Kujala/ Anterior knee pain scale (AKPS) | 12th sessions for four weeks, ,outcome measures will take place both, at the baseline when intervention start and four weeks, following the intervention
  we will use the Kujala scale to measure functional limitations, a reliable instrument retest reliability of 0.9 in patient with PFPS, total 13 self-reported questionnaire. AKPS graded 0 to 100, 100 being the highest possible score with no pain and disability. Lower scores reflect greater pain and disability.

CONTACTS AND LOCATIONS:
Locations (1):
- Saddar, Karachi, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Efficacy of electromyographic-biofeedback supplementation training with patellar taping on quadriceps strengthening in patellofemoral pain syndrome among young adult male athletes — https://pubmed.ncbi.nlm.nih.gov/33922866/
- See also: McConnell patellar taping on postural control of women with patellofemoral pain syndrome — https://www.researchgate.net/publication/343197750_McConnell_patellar_taping_on_postural_control_of_women_with_patellofemoral_pain_syndrome_randomized_clinical_trial